CLINICAL TRIAL: NCT01431066
Title: Continuous Low Energy Pulsed Radio Frequency Electromagnetic Field Therapy for the Treatment of Plantar Fasciopathy
Brief Title: ActiPatch Plantar Fasciitis Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: BioElectronics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H11-01828
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2011-09

CONDITIONS: Plantar Fasciitis; Plantar Fasciopathy
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Sham device that resembles the Actipatch PRFE device, including the light that illuminates when active, but the transmitting function has been disabled.
  Interventions: Device: Sham pulsed radio-frequency electromagnetic device
- Actipatch (Experimental): Use of the Actipatch PRFE device that is integrated into a viscoelastic heel pad for the treatment of plantar fasciopathy
  Interventions: Device: ActiPatch PRFE Device

INTERVENTIONS:
Device: Sham pulsed radio-frequency electromagnetic device — Disabled PRFE device
  Arms: Control
Device: ActiPatch PRFE Device — Actipatch PRFE device
  Arms: Actipatch

SUMMARY:
Plantar fasciopathy is a chronic condition affecting both sedentary populations, individuals in the workplace who must stand for prolonged periods of time, and athletes. It can be disabling. There is no single accepted treatment course that is recommended in the literature.

The use of pulsed radio-frequency electromagnetic (PRFE) devices has been proposed as a treatment option in chronic soft-tissue injury due to its ability to reduce pain and inflammation.

The proposed study will investigate the efficacy of the use of a PRFE device for the treatment of chronic heel pain using a double blind randomized placebo controlled design study.

ELIGIBILITY:
Inclusion Criteria:

* All patients with diagnosis of plantar fasciitis agreeing to participate
* Over 18 years old
* Able to wear unit and keep data up-to-date records of use
* Agree to forgo additional treatments during the study period

Exclusion Criteria:

* Patients who have refused, are unable to give or have withdrawn consent
* Patients with heel pain present less than 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for pain | 4 Weeks Follow-up

SECONDARY OUTCOMES:
Visual analog scale for pain | 26 weeks
Foot and ankle disability index | 26 weeks
Tegner activity scale | 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Medicine, Vancouver, British Columbia, Canada